CLINICAL TRIAL: NCT05632848
Title: The Efficacy and Safety of Chidamide Combined With Zimberelimab in the Treatment of Metastatic Triple-negative Breast Cancer Patients: A Single-armed, Phase II Trial
Brief Title: Chidamide Combined With Zimberelimab in the Treatment of Metastatic Triple-negative Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC 019
Record Dates: First submitted 2022-11-06; First posted 2022-12-01 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-07

CONDITIONS: Triple Negative Breast Cancer
Keywords: Chidamide plus Zimberelimab
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — zimberelimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Chidamide and Zimberelimab
  Interventions: Drug: Chidamide combined with Zimberelimab

INTERVENTIONS:
Drug: Chidamide combined with Zimberelimab — Chidamide: 30mg each time, orally, biw; Zimberelimab, 240mg, IV, every 3 weeks.
  Other Names: Chidamide (Tucidinostat)

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of a new treatment regimen (Chidamide combined with Zimberelimab) in the treatment of patients with metastatic triple negative breast cancer after the second-line therapy.

DETAILED DESCRIPTION:
This is a phase II, single center, prospective, single arm clinical trial. The objective of the study is to evaluate the efficacy and safety of a new treatment regimen (Chidamide combined with Zimberelimab) in the treatment of patients with metastatic triple negative breast cancer after the second-line therapy. This study plans to recruit 47 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of triple-negative breast cancer on primary tumour at diagnosis/on biopsy of metastasis.
* At least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Fail first-line or above anti-tumor treatment.
* Adequate organ function including bone marrow, renal function, hepatic function, and cardiac reserve.
* Compliance with the study protocol.
* Have provided written and signed informed consent.
* Minimum life expectancy 16 weeks.

Exclusion Criteria:

* Pregnant or breast feeding.
* Uncontrolled medical problems.
* Evidence of active acute or chronic infection.
* Hepatic, renal, cardiac, or bone marrow dysfunction.
* Concurrent malignancy or history of other malignancy within the last five years.
* Known severe hypersensitivity to Chidamide or Zimberelimab
* Patients were unable or unwilling to comply with program requirements.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 18 months
  The proportion of patients with measurable tumor size reduction of a predefined amount (complete response [CR], partial response [PR]) according to the response evaluation criteria in solid tumors (RECIST) version 1.1. Complete Response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm (<1 cm). Partial Response: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | 18 months
  The proportion of patients with measurable tumor size stable lasting ≥24 weeks (stable disease [SD]) or its size reduction of a predefined amount (complete response [CR], partial response [PR]) following the response evaluation criteria in solid tumors (RECIST) version 1.1. Complete Response (CR) and Partial Response (PR) are defined in Primary Outcome Measure. Stable Disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (progressive disease), taking as reference the smallest sum diameters while on study. Progressive Disease: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (0.5 cm). (Note: the appearance of one or more new lesions is also considered progression).
Progression Free Survival (PFS) | 24 months
  The interval time from the date of initiation treatment for metastatic breast cancer to the date of the first documented disease progression or death due to any cause.
Overall Survival (OS) | 30 months
  The interval time from the date of initiation treatment for metastatic breast cancer to the date of death from any cause.
Occurrence and severity of AEs | 30 months
  Occurrence and severity of AEs by NCI-CTCAE v5. Changes in laboratory parameters (hematology and serum chemistry), vital signs and ECG parameters. Grade 3 or 4 abnormalities in serum chemistry laboratory parameters.

OTHER OUTCOMES:
Biomarkers related to efficacy | 24 months
  Baseline tumor biopsy from metastatic or recurrent lesions was required, we analyze and compare the difference of tumor immune microenvironment among patients with different responses to this intervention via the single cell sequencing of acquired tumor biopsy.
  And peripheral blood samples were collected at baseline, one day before the second cycle treatment and the date of withdrawal from this clinical trial confirmed by researchers. Then peripheral blood mononuclear cell cluster analysis will be performed and compared their changes before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-yu Yuan, M.D., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong, China